CLINICAL TRIAL: NCT02494791
Title: Universal Screening for Lynch Syndrome in Women With Endometrial and Non-Serous Ovarian Cancer
Acronym: LS2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Health Network, Toronto (Other)
Collaborators: Mount Sinai Hospital, Canada (Other); Sunnybrook Health Sciences Centre (Other); Hamilton Health Sciences Corporation (Other); Toronto Metropolitan University (Other); University of Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 14-8533CE
Record Dates: First submitted 2015-07-07; First posted 2015-07-10 (Estimated); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Lynch Syndrome; Endometrial Neoplasms; Ovarian Neoplasms; Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms, Hereditary Nonpolyposis; Endometrial Neoplasms; Ovarian Neoplasms; Colorectal Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Endometrial and Ovarian Cancer Participants (Other): All study subjects will be offered the same options for screening and follow-up.
  Interventions: Behavioral: Questionnaire, Educational Material

INTERVENTIONS:
Behavioral: Questionnaire, Educational Material — Participants in this study will be given educational material about Lynch Syndrome and genetic testing for this condition. They will be asked to complete questionnaires about their family cancer history, personal health history and attitudes toward genetic testing.

SUMMARY:
This study will maximize identification of women with Lynch Syndrome using an enhanced screening strategy to identify those at risk. These women will be referred to genetic counselling for testing and those found to have Lynch Syndrome will be asked to invite first degree relatives to participate and undergo genetic testing for Lynch Syndrome. Screening guidelines and risk reducing surgery options for participants found to have Lynch Syndrome will be reinforced by the study and adherence to these guidelines will be assessed annually for ten years following Lynch Syndrome diagnosis to assess the impact and cost-effectiveness of this enhanced screening approach.

DETAILED DESCRIPTION:
Lynch Syndrome increases an individual's risk for several cancers, such as colorectal, endometrial (EC) and certain types of ovarian cancer (OC). Lynch Syndrome is caused by inherited changes in mismatch repair (MMR) genes. In this study we will establish the proportion of EC and OC patients with Lynch Syndrome. We will screen all EC and OC patients by performing MMR immunohistochemistry (IHC) on their surgical specimen. These data will then be used along with family history data to determine which women are at high risk of Lynch Syndrome. We will facilitate the referral of all women at risk for Lynch Syndrome to genetic counselling on behalf of their treating physician. First degree relatives of those patients found to have Lynch Syndrome who consent to participate in the study will also be referred to genetics by the study PI. We will encourage all participants found to have Lynch Syndrome to attend regular colonoscopy screening to prevent colorectal cancer, and (for females with Lynch Syndrome) consideration of gynecologic risk reducing surgery to prevent endometrial and ovarian cancers. We will assess adherence to Lynch Syndrome screening guidelines in this population and will determine if our universal screening strategy is feasible and cost-effective for widespread implementation across Canada in an effort to prevent Lynch Syndrome associated cancers in women and their families. In addition to this, consenting patients may provide blood and tumour tissue samples for sequencing studies which will investigate the genetic basis for Lynch Syndrome and shed light on cases of MMR loss in the absence of germline mutation.

ELIGIBILITY:
Inclusion Criteria (Patients):

* 18-70 years old
* endometrial cancer (all grades, stages and histologic subtypes except stromal sarcoma, carcinosarcoma)
* cancer diagnosed within 6 months of consent
* tumour tissue available for MMR IHC
* willing and able to give informed consent for participation in study

Exclusion Criteria (Patients):

* patients under 18 years old or over 70 years old
* patients with uterine adenosarcoma, leiomyosarcoma or endometrial stromal sarcoma
* patients with pure serous or pure mucinous ovarian carcinoma
* patients unwilling or unable to participate in the informed consent process

Inclusion Criteria (First-degree Relatives)

* minimum 18 years old
* reside in Canada
* willing and able to give informed consent for participation in study

Exclusion Criteria (First-degree Relatives):

* under 18 years old
* reside outside of Canada
* unwilling or unable to participate in the informed consent process

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 886 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2020-07 (Actual); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Adherence to screening guidelines (colonoscopy and gynecologic risk-reducing surgery) in participants found to have Lynch Syndrome | short-term assessment at 1 year after diagnosis, long-term assessment for up to 10 years after diagnosis
  Participants found to have Lynch Syndrome will be followed after diagnosis and asked to update the study annually with information about any colorectal cancer screening (colonoscopy) and/or gynecologic risk-reducing surgery they've undergone. This information will be used to assess the success of the enhanced universal screening protocol in helping treat pre-cancerous lesions and therefore prevent a possible cancer as well as aid in detection of early malignancies that otherwise may have gone undetected.
Cost-effectiveness of universal enhanced screening strategy to identify women with Lynch Syndrome and their family members via cascade testing | short-term assessment at 1 year after diagnosis, long-term assessment for up to 10 years after diagnosis
  Data about adherence to screening guidelines and the outcome of screening procedures will be used to inform cost-effectiveness models assessing the feasibility of implementing this enhanced universal screening strategy for Lynch Syndrome in institutions across Canada.

SECONDARY OUTCOMES:
Incidence of Lynch Syndrome in an unselected group of women with endometrial and non-serous ovarian cancer | 3 years
  This study will add data about the number of Lynch Syndrome cases among a large cohort of endometrial cancer patients in Canada, adding to previous work. This will be the first prospective study to assess Lynch Syndrome incidence in non-serous, non-mucinous ovarian cancer patients in Canada.
Discovery of novel genetic mutations and molecular events in unexplained MMR loss (Lynch-like Syndrome) | 3-5 years
  This study will investigate tumour samples from women with unexplained MMR loss (MMR IHC deficient without a germline mutation) to probe what other factors may contribute to Lynch-like Syndrome. Currently these patients are believed to have an intermediate risk for Lynch-associated cancers and are counselled accordingly. Further investigation into the biology of this condition may yield more effective strategies for stratifying and managing risk for Lynch-like Syndrome patients.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Ferguson, MD, Principal Investigator — Princess Margaret Cancer Centre
Locations (1):
- University Health Network - Princess Margaret Hospital, Toronto, Ontario, Canada